CLINICAL TRIAL: NCT05417711
Title: Efficacy of Transcutaneous Vagus Nerve Stimulation Paired With Tailor-Made Notched Music Therapy Versus Tailor-made Notched Music Training for Chronic Subjective Tinnitus: A Multicenter, Randomized, Double-blind, Controlled Clinical Trial
Brief Title: Efficacy of Transcutaneous Vagus Nerve Stimulation Paired With Tailor-Made Notched Music Therapy Versus Tailor-made Notched Music Training for Chronic Subjective Tinnitus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Zhongshan People's Hospital, Guangdong, China (Other); Affiliated Zhuhai Hospital of Southern Medical University (Unknown); Guangzhou Panyu Central Hospital (Other); Shenshan Medical Center, Memorial Hospital of Sun Yat-sen University (Unknown); Eighth Affiliated Hospital, Sun Yat-sen University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Southern Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-KY-074
Record Dates: First submitted 2022-06-06; First posted 2022-06-14 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Tinnitus, Subjective; Vagus Nerve Stimulation; Music Therapy; Double-Blind Method; Female; Male; Humans; Treatment Outcome
Keywords: Chronic subjective tinnitus; Tailor-made notched music training; Vagus nerve stimulation; Electroencephalogram; Clinical trial
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: The subjects included in the study are randomized by a unified randomization center. The randomization center will number the subjects with the random number table generated by the computer, and then arrange them in the order of number. The subjects will be randomly divided into groups in turn, and the subjects in the groups will be numbered with the random number table. The first half of the subjects with a larger number in the groups will be divided into the experimental group (tVNS paired with TMNMT), and the rest into the control group (TMNMT).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the whole clinical research process, the subjects and researchers participating in the efficacy and safety evaluation should be in a blind state, that is, neither of them knows the specific intervention measures given to the subjects. For participant, the treatment equipment is exactly the same between the two groups. Also, 10 seconds sham stimulation at the beginning of treatment is set in the control group for minimizing risk of participants being able to guess treatment allocation. The randomized allocation is completed by a unified randomization center. Therefore, the investigators in each center just know "A" or "B" for the allocation information of each participant. For outcomes assessors, they are only responsible for baseline and follow-up assessment during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Vagus Nerve Stimulation Paired with Tailor-Made Notched Music Therapy (Experimental): The participants receive 30 minutes / time, 4 times / day, continuous 3 months of auditory tVNS combined with TMNMT. The stimulation intensity used in each course was set to the highest level that the patient could tolerate. The participants listen to the tailor-made notched music at the same time.
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation Paired with Tailor-Made Notched Music Therapy
- Tailor-made Notched Music Training (Active Comparator): Similarly, 30 minutes / time, 4 times / day, continuous 3 months of TMNMT is received every day. The setting of parameters and the selection of music were the same as those in the experimental group. At the beginning of TMNMT, 10 s of sham stimulation set according to the standard of the experimental group is given.
  Interventions: Device: Tailor-made Notched Music Training

INTERVENTIONS:
Device: Transcutaneous Vagus Nerve Stimulation Paired with Tailor-Made Notched Music Therapy — The pulse frequency of vagus nerve stimulation is 25 Hz, the pulse width is 200 US, and the intensity is 1-10 mA. Tailor-made notched music is produced by filtering a frequency band of 1/2 octave width centered at the individual tinnitus frequency. When two sides of tinnitus frequencies are different, each side of music are filtered respectively, according to the different tinnitus frequency. When only have unilateral tinnitus or bilateral tinnitus in the same central frequency, both sides of music are filtered with the same tinnitus frequency. The tVNS and TMNM begin at the same time during treatment.
  Arms: Transcutaneous Vagus Nerve Stimulation Paired with Tailor-Made Notched Music Therapy
Device: Tailor-made Notched Music Training — Tailor-made notched music is produced by filtering a frequency band of 1/2 octave width centered at the individual tinnitus frequency. When two sides of tinnitus frequencies are different, each side of music are filtered respectively, according to the different tinnitus frequency. When only have unilateral tinnitus or bilateral tinnitus in the same central frequency, both sides of music are filtered with the same tinnitus frequency. At the beginning of TMNMT, 10 seconds sham vagus nerve stimulation is output, whose parameters are as same as experimental group.
  Arms: Tailor-made Notched Music Training

SUMMARY:
This clinical study is a prospective, multicenter, randomized, controlled, double-blind clinical study. Sun Yat Sen Memorial Hospital of Sun Yat sen University was the central unit, and Nanjing First Hospital, Sun Yat Sen people's Hospital, Guanfzhou Panyu central Hospital and Zhuhai integrated traditional Chinese and Western medicine hospital were the cooperative units. In this study, 388 patients with chronic subjective tinnitus were recruited. In view of chronic subjective tinnitus, a common ear disease, the study gave the patients three months of treatment with transcutaneous vagus nerve stimulation paired with tailor-made notched music therapy or tailor-made notched music training alone. By comparing the changes of subjective scale scores related to tinnitus before and after treatment in patients receiving two different therapies, such as THI, VAS, BAI, BDI, PSQI, to evaluate the efficacy of the two therapies, so as to judge whether transcutaneous vagus nerve stimulation paired with tailor-made notched music therapy is better than tailor-made notched music training alone. In addition, the study will continue to follow up the patients after the treatment for one year to observe the difference in the long-term sustained efficacy of the two therapies. This clinical study will also evaluate the two therapies from the perspective of compliance and safety, and explore the factors that affect the efficacy of the two therapies.

DETAILED DESCRIPTION:
Unified rules for filling in case report forms：

* All case report forms must be completed by designated and trained researchers.
* Two data managers independently input and proofread the data in duplicate.
* The data manager will modify, confirm and enter the data according to the scales written by participant.
* The locked data file will not be changed.
* Use medical terms / concepts to record AES . The type, degree, occurrence time, duration, treatment measures and treatment process shall be recorded in detail.

Sample size estimation:

* △ THI≥ 7 points in the comparison between groups indicates that the difference in efficacy has clinical significance, the superiority margin is established.
* The pre-test results showed that △ THI = -10.2 points, SD = 10.0 points in the two groups after the treatment.
* According to unilateral inspection standard α= 0.025, inspection efficacy 1- β= 0.80, using two sample t-test to estimate the sample size, the results show that at least 155 subjects are included in each group.
* Further estimation was made according to the loss of follow-up rate of 20%. Finally, at least 194 subjects (388 persons in total) should be included in each group.
* PASS 21.0.03 (NCSs, LLC, Kaysville, Utah, USA) is adopted for the above calculation.

Plan for missing data：

* If the subject uses the drugs, treatment or surgery prohibited in the protocol, the subject will no longer meet the conditions of the clinical study and will be deemed to have withdrawn from the study.
* If the event occurs before 3 months of treatment, the subject's data will no longer be used for statistical analysis of subsequent data.
* If the event occurs in the follow-up period after the completion of treatment, the data of the subject before and after treatment shall be retained. The data in the follow-up period shall be regarded as missing data and filled with corresponding methods for full analysis set analysis.
* For the missing data caused by the loss of follow-up, this study will use the method of multiple imputation to estimate the missing value.
* The research subjects who failed in screening will provide corresponding treatment according to their own conditions and clinical guidelines. These subjects will not be included in the clinical study.

Statistical analysis plan:

When considering the influence of baseline, the continuous variables were analyzed by covariance analysis, and the qualitative indicators were tested by CMH test or logistic regression.

Primary analysis： Using covariance analysis to compare the different changes of THI scores between two groups after 3-month treatment, controlled for age and baseline THI.

Secondary analysis： Using covariance analysis to compare the different changes of VAS, BAI, BDI, PSQI scores between two groups after 3-month treatment, controlled for age and baseline values corresponding to each scale.

Using a repeated measure ANOVA to compare the different changes of THI, VAS, BAI, BDI, PSQI between two groups at 3, 6 and 12 follow-up visits.

Using Chi square test or Fisher exact test to compare the different efficient rate between two groups after 3-month treatment.

Exploratory analysis:

Using multiple linear regression analysis to explore the factors affecting the short-term and long -term efficacy of the two treatments, such as age, hearing loss threshold, tinnitus loudness, tinnitus frequency and so on.

Using Independent two sample t-test or nonparametric analysis to compare the differences in EEG- or fMRI-related indicators between two groups.

Safety analysis:

Using Pearson's chi-square test to compare the difference of adverse event incidence rate between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tinnitus as the main complaint: the patients subjectively feel the sound in the ear or deep part of the head without internal or external sound stimulation, and therefore seek medical treatment
* Chronic (≥ 6 months) and tonal tinnitus
* Age 18-60
* Tinnitus frequency is 125-8000 Hz
* Hearing threshold at each frequency shall not exceed 70 dB HL

Exclusion Criteria:

* Patients with conductive deafness, history of middle ear surgery, pulsatile tinnitus caused by vascular distortion and tinnitus caused by Meniere disease
* History of head trauma, central nervous system diseases, mental diseases and drug abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 388 (Estimated)
Dates: Start 2023-11-23 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Tinnitus Handicap Inventory (THI) scores for short-term efficacy assessment | From baseline to 3-month follow-up visit
  Difference in the change of THI scores between two groups after 3-month treatment. The THI evaluates the severity of tinnitus in terms of emotion and function. The global scores of THI range from 0 (no disability) to 100 (serve disability).

SECONDARY OUTCOMES:
Changes in scores of Visual Analog Scale (VAS) for short-term efficacy assessment | From baseline to 3-month follow-up visit
  Difference in the change of VAS scores between two groups after 3-month treatment. The total VAS scores range from 0 (negligible) to 10 (too nosiy to tolerate), reflecting the loudness of tinnitus patients feel.
Changes in scores of Beck Anxiety Inventory (BAI) for short-term efficacy assessment | From baseline to 3-month follow-up visit
  Difference in the change of BAI scores between two groups after 3-month treatment. The total BAI scores range from 0 (normal) to 63 (serve anxiety), reflecting the degree of anxiety.
Changes in scores of Beck Depression Inventory (BDI) for short-term efficacy assessment | From baseline to 3-month follow-up visit
  Difference in the change of BDI scores between two groups after 3-month treatment. The total BDI scores range from 0 (normal) to 63 (serve depression), reflecting the degree of depression.
Changes in scores of Pittsburgh sleep quality index (PSQI) for short-term efficacy assessment | From baseline to 3-month follow-up visit
  Difference in the change of PSQI scores between two groups after 3-month treatment. The total PSQI scores range from 0 (sleep well) to 21 (quite poor sleep), reflecting the sleep quality.
Changes of Tinnitus Handicap Inventory (THI) scores in the two groups for long-term efficacy assessment | From 3-month follow-up visit to 12-month follow-up visit
  Difference in changes of THI between two groups from 3-month follow-up visit to 12-month follow-up visit. The THI evaluates the severity of tinnitus in terms of emotion and function. The global scores of THI range from 0 (no disability) to 100 (serve disability).
Changes of Visual Analog Scale (VAS) scores in the two groups for long-term efficacy assessment | From 3-month follow-up visit to 12-month follow-up visit
  Difference in changes of VAS between two groups from 3-month follow-up visit to 12-month follow-up visit. The total VAS scores range from 0 (negligible) to 10 (too nosiy to tolerate), reflecting the loudness of tinnitus patients feel.
Changes of Beck Anxiety Inventory (BAI) scores in the two groups for long-term efficacy assessment | From 3-month follow-up visit to 12-month follow-up visit
  Difference in changes of BAI between two groups from 3-month follow-up visit to 12-month follow-up visit. The total BAI scores range from 0 (normal) to 63 (serve anxiety), reflecting the degree of anxiety.
Changes of Beck Depression Inventory (BDI) scores in the two groups for long-term efficacy assessment | From 3-month follow-up visit to 12-month follow-up visit
  Difference in changes of PSQI between two groups from 3-month follow-up visit to 12-month follow-up visit. The total BDI scores range from 0 (normal) to 63 (serve depression), reflecting the degree of depression.
Changes of Pittsburgh sleep quality index (PSQI) scores in the two groups for long-term efficacy assessment | From 3-month follow-up visit to 12-month follow-up visit
  Difference in changes of PSQI between two groups from 3-month follow-up visit to 12-month follow-up visit. The total PSQI scores range from 0 (sleep well) to 21 (quite poor sleep), reflecting the sleep quality.
The effective rate of relieving chronic subjective tinnitus in the two groups | From baseline to 3-month follow-up visit
  Group effective rate = number of patients in each group who completed 3 months of treatment and whose THI score decreased by ≥ 7 points / number of patients in each group who completed 3 months of treatment.
The difference of functional connectivity based on resting state electroencephalogram (EEG) between the two groups | From baseline to 12-month follow-up visit
  The difference of functional connectivity based on resting state electroencephalogram (EEG) in the two groups from baseline to 12-month follow-up visit. The functional connectivity is defined as the correlation between two different brain regions based on coherence or phase synchronization.
The difference of effective connectivity based on resting state electroencephalogram (EEG) between the two groups | From baseline to 12-month follow-up visit
  The difference of effective connectivity based on resting state electroencephalogram (EEG) in the two groups from baseline to 12-month follow-up visit. The effective connectivity is defined as the directed functional connectivity between two brain regions based on granger causality analysis.
The difference of functional connectivity based on functional magnetic resonance imaging (fMRI) between the two groups | From baseline to 12-month follow-up visit
  The difference of functional connectivity based on functional magnetic resonance imaging (fMRI) in the two groups from baseline to 12-month follow-up visit. The functional connectivity is defined as the Pearson's correlation between two different brain regions.
The difference of effective connectivity based on functional magnetic resonance imaging (fMRI) between the two groups | From baseline to 12-month follow-up visit
  The difference of effective connectivity based on functional magnetic resonance imaging (fMRI) in the two groups from baseline to 12-month follow-up visit. The effective connectivity is defined as the directed functional connectivity between two brain regions based on granger causality analysis.

OTHER OUTCOMES:
Incidence of treatment-related adverse events | From baseline to 12-month follow-up visit
  Treatment related adverse events in two groups include: auditory system related adverse reactions caused by treatment, such as auricle burn, earache, hearing loss, tinnitus aggravation, and head injury Dizziness, headache, palpitation, vomiting and other non auditory system related adverse reactions. Incidence of adverse events = number of treatment-related adverse events during treatment / total number of participants in treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yuexin Cai Cai, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

REFERENCES:
- [Background] Piccirillo JF, Rodebaugh TL, Lenze EJ. Tinnitus. JAMA. 2020 Apr 21;323(15):1497-1498. doi: 10.1001/jama.2020.0697. No abstract available. PMID 32176246
- [Background] Stockdale D, McFerran D, Brazier P, Pritchard C, Kay T, Dowrick C, Hoare DJ. An economic evaluation of the healthcare cost of tinnitus management in the UK. BMC Health Serv Res. 2017 Aug 22;17(1):577. doi: 10.1186/s12913-017-2527-2. PMID 28830503
- [Background] Henry JA, Reavis KM, Griest SE, Thielman EJ, Theodoroff SM, Grush LD, Carlson KF. Tinnitus: An Epidemiologic Perspective. Otolaryngol Clin North Am. 2020 Aug;53(4):481-499. doi: 10.1016/j.otc.2020.03.002. Epub 2020 Apr 30. PMID 32362561
- [Background] Langguth B, Elgoyhen AB, Cederroth CR. Therapeutic Approaches to the Treatment of Tinnitus. Annu Rev Pharmacol Toxicol. 2019 Jan 6;59:291-313. doi: 10.1146/annurev-pharmtox-010818-021556. Epub 2018 Jul 25. PMID 30044727
- [Background] 龚树生 贺 王. 解读美国《耳鸣临床应用指南》 [J]. 中华耳科学杂志, 2016, 14(2): 4
- [Background] Stein A, Engell A, Junghoefer M, Wunderlich R, Lau P, Wollbrink A, Rudack C, Pantev C. Inhibition-induced plasticity in tinnitus patients after repetitive exposure to tailor-made notched music. Clin Neurophysiol. 2015 May;126(5):1007-15. doi: 10.1016/j.clinph.2014.08.017. Epub 2014 Sep 6. PMID 25441152
- [Background] Okamoto H, Stracke H, Stoll W, Pantev C. Listening to tailor-made notched music reduces tinnitus loudness and tinnitus-related auditory cortex activity. Proc Natl Acad Sci U S A. 2010 Jan 19;107(3):1207-10. doi: 10.1073/pnas.0911268107. Epub 2009 Dec 28. PMID 20080545
- [Background] Tyler R, Cacace A, Stocking C, Tarver B, Engineer N, Martin J, Deshpande A, Stecker N, Pereira M, Kilgard M, Burress C, Pierce D, Rennaker R, Vanneste S. Vagus Nerve Stimulation Paired with Tones for the Treatment of Tinnitus: A Prospective Randomized Double-blind Controlled Pilot Study in Humans. Sci Rep. 2017 Sep 20;7(1):11960. doi: 10.1038/s41598-017-12178-w. PMID 28931943
- [Background] Rammo R, Ali R, Pabaney A, Seidman M, Schwalb J. Surgical Neuromodulation of Tinnitus: A Review of Current Therapies and Future Applications. Neuromodulation. 2019 Jun;22(4):380-387. doi: 10.1111/ner.12793. Epub 2018 Jul 17. PMID 30015361
- [Background] Clancy JA, Mary DA, Witte KK, Greenwood JP, Deuchars SA, Deuchars J. Non-invasive vagus nerve stimulation in healthy humans reduces sympathetic nerve activity. Brain Stimul. 2014 Nov-Dec;7(6):871-7. doi: 10.1016/j.brs.2014.07.031. Epub 2014 Jul 16. PMID 25164906
- [Background] Yap JYY, Keatch C, Lambert E, Woods W, Stoddart PR, Kameneva T. Critical Review of Transcutaneous Vagus Nerve Stimulation: Challenges for Translation to Clinical Practice. Front Neurosci. 2020 Apr 28;14:284. doi: 10.3389/fnins.2020.00284. eCollection 2020. PMID 32410932
- [Background] 曾祥丽, 郑可, 岑锦添, et al. 经皮耳迷走神经刺激治疗慢性耳鸣的疗效观察 [J]. 临床耳 鼻咽喉头颈外科杂志, 2021, 35(02): 105-8.
- [Background] Shim HJ, Kwak MY, An YH, Kim DH, Kim YJ, Kim HJ. Feasibility and Safety of Transcutaneous Vagus Nerve Stimulation Paired with Notched Music Therapy for the Treatment of Chronic Tinnitus. J Audiol Otol. 2015 Dec;19(3):159-67. doi: 10.7874/jao.2015.19.3.159. Epub 2015 Dec 18. PMID 26771015
- [Background] Yakunina N, Nam EC. Direct and Transcutaneous Vagus Nerve Stimulation for Treatment of Tinnitus: A Scoping Review. Front Neurosci. 2021 May 28;15:680590. doi: 10.3389/fnins.2021.680590. eCollection 2021. PMID 34122002
- [Background] Stein A, Wunderlich R, Lau P, Engell A, Wollbrink A, Shaykevich A, Kuhn JT, Holling H, Rudack C, Pantev C. Clinical trial on tonal tinnitus with tailor-made notched music training. BMC Neurol. 2016 Mar 17;16:38. doi: 10.1186/s12883-016-0558-7. PMID 26987755
- [Background] 蔡跃新, 孙映凤, 杨海弟, et al. 个性化切迹音乐治疗主观性耳鸣的初步观察 [J]. 中华耳科学杂志, 2017, 15(04): 465-70.